CLINICAL TRIAL: NCT03733288
Title: Outcome, Process and Economic Evaluation of a Randomised Controlled Trial to Reduce Call Agents' Sitting Time at Work: Project SLAMM
Brief Title: Reducing Contact Centre Call Agents' Sitting Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: University of Liverpool (Other); University of Leicester (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Lee Graves, Senior Lecturer, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-SPS-Graves1
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Sedentary Lifestyle; Physical Activity
Keywords: Intervention; Workplace; Sedentary behaviour; Physical activity; Adults; Economic; Evaluation
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLAMM (Experimental): Multi-component intervention (Education and training sessions, Support emails, Team leader training)
  Interventions: Behavioral: Education and training sessions; Behavioral: Support emails; Behavioral: Team leader training
- SLAMM+ (Experimental): Multi-component intervention (Education and training sessions, Support emails, Team leader training, Height-adjustable workstation)
  Interventions: Behavioral: Education and training sessions; Behavioral: Support emails; Behavioral: Team leader training; Device: Height-adjustable workstation

INTERVENTIONS:
Behavioral: Education and training sessions — Agents will be invited to attend sessions in intervention week 1, 3, 9, and month 6. Sessions will introduce (week 1) and reinforce (week 3, 9, month 6) the intervention aims, benefits of and ways to move more and sit less, with emphasis on active breaks. Feedback from baseline assessment will be provided and discussed in week 3 (health data) and 9 (activity data) and month 6 (health and activity data from the 12-week assessment). Each session will include discussion of daily standing/walking goals set by the research team, with timers and a goal log provided to participants in week 1 to enable self-monitoring. The Stand Up champions, and their role to encourage daily movement and sitting reduction through modelling and verbal support, will be communicated and reinforced in each session.
Behavioral: Support emails — Agents will receive support emails weekly (weeks 1-12) then monthly (months 4-9) across the intervention. Each email includes an infographic that encourages moving more and sitting less at work.
Behavioral: Team leader training — Team leaders in the participating organisation will be invited to attend a training session before the intervention starts. The training aims to enhance team leader's capabilities to demonstrate positive movement and sitting behaviours at work and promote call agents to sit less and move more at work. Team leaders will be asked to include the intervention as an agenda item in their weekly team meetings with their call agents and their 1:1 sessions with call agents. Team leaders will be encouraged to incorporate walking into their 1:1 meetings with call agents.
Device: Height-adjustable workstation — After baseline, agents in the SLAMM+ arm will have a height-adjustable workstation installed on their existing workplace desk. This will enable work in a seated or standing position, with flexibility to alternate between postures. Desk installation will occur with support from the onsite organisation health and safety team. The research team will brief participants on safe and effective workstation use. A laminated sheet will be fixed to each workstation to remind participants of safe and effective use.
  Arms: SLAMM+

SUMMARY:
The study investigates whether a workplace intervention can encourage highly sedentary contact centre call agents to sit less and move more at work. The effect of the intervention will be assessed at 12 weeks and 9 months. The hypothesis is that the intervention will reduce workplace sitting and increase workplace standing and light walking.

DETAILED DESCRIPTION:
Study Design:

This randomised controlled trial has two experimental treatment arms, SLAMM and SLAMM+.

Recruitment:

- Organisation Level:

Organisation recruitment is via a tender process. A recruitment infographic and application form will be emailed to contact centres affiliated with the Call North West Forum (~700 centres in the North West of England). Organisations have 3-weeks to apply by submitting the application form to the research team. Applications will be reviewed and ranked, and if multiple suitable organisations apply, a meeting will be held with each organisation to discuss the organisation's suitability. Applicants will be notified of the decision via telephone call and subsequent confirmation email, with feedback as to why they were unsuccessful (if applicable). The gatekeeper from the successful organisation will receive a gatekeeper participant information and consent form to sign prior to individual level recruitment.

- Individual Level

Call Agents: Study information sessions during work hours at the organisation, and an email containing a participant information sheet, will be used to recruit call agents. Agents have 2 weeks to express interest. Interested employees will be screened for eligibility using stated criteria via telephone or in person. If inclusion criteria are met, written informed consent will be obtained and baseline assessments scheduled. There will be no racial or gender bias in participant selection.

Stand Up Champions: During agent recruitment, agents will be told about the opportunity to be a stand up champion and have 2 weeks to express interest. There is no limit to the number of champions recruited.

Team Leaders and Management: A participant information sheet and consent form sent via email will be used to recruit team leaders (focus group), middle managers (focus group) and senior managers (interviews) for the process evaluation on intervention acceptability and feasibility at 12 weeks and 9 months.

Group Assignment:

Following baseline data collection, randomisation to the SLAMM or SLAMM+ arm will occur using a number generator by a member of the research team not involved in recruitment. The unit of randomisation will be at the individual level. The participants will be informed of the outcome of the randomisation via email.

Data Collection:

Participants will complete assessments at baseline, 12-weeks and 9 months. Individual assessments include surveys, cardiometabolic and anthropometric measures, and objective physical activity and sedentary behaviour monitoring. Individual assessments will take place within the participant's work site during work hours. Participants will be asked to fast for a minimum of 8 hours, avoid smoking and active transport on the morning of the assessment, avoid alcohol, tea or coffee intake for a minimum of 12-h prior to assessments, and avoid strenuous exercise for a minimum of 24-h prior to assessments. A sub-sample of participants from each treatment arm will be randomly selected to take part in focus groups at 12 weeks and 9 months to evaluate intervention acceptability and feasibility.

Sample Size:

Allowing for moderate drop out, the study aimed to recruit 30 participants per arm and retain 23 participants per arm. A sample size of 23 per arm would achieve 90% power (alpha 5%; two-tailed) to detect a minimum difference of 60 minutes/8-hour workday between arms for workplace sitting time (primary outcome: expected standard deviation of 60 minutes/day).

Analyses:

- Outcome evaluation:

Data will be analysed by an independent statistician (blinded to the treatment arms) using STATA (STATACorp LP) with the alpha level set at p≤0.05. For continuous outcomes, intervention effects and changes within groups will be estimated using linear mixed models. Models will include fixed terms for group (intervention 1/intervention 2), time (3 or 9 months), and group-time interaction, with potential confounders. Estimates of changes within groups, and differences between groups, will be obtained using marginal means and pairwise comparisons of marginal means of the outcome.

- Process evaluation:

Inductive thematic analysis will identify, analyse and explore themes from focus group and interview data on intervention acceptability and feasibility at 12 weeks and 9 months. Surveys will also assess intervention acceptability and feasibility at 12 weeks and 9 months.

- Economic evaluation:

The economic evaluation will be conducted from three perspectives. From the health sector perspective, trial-and model-based cost-utility analyses will be performed to show the cost of the intervention per quality adjusted life year. From the employer perspective, a cost-effectiveness analysis will be conducted to show the cost of the intervention per change in productivity. From the broader societal perspective, a cost-consequence analysis will be presented outlining all the costs and effects (in their natural units) which are incurred by the various stakeholders including the participants, and the participant's family and friends.

ELIGIBILITY:
Call agents inclusion criteria:

* Full time member of staff (≥0.6 full time or part time equivalent worker in a permanent or temporary/agency position)
* Call agent job role
* Based onsite throughout the trial period
* Access to a work telephone and desktop computer with internet
* Ambulatory

Call agents exclusion criteria:

* Health problems that would impact ability to stand for 10 minutes at a time
* Planned absence >3 weeks during first 3 months of the trial
* Planned relocation to another workplace/site during the first 3 months of the intervention
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Change in workplace sitting time at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  An activpal monitor will objectively assess habitual sitting time for 24 hours over 7 consecutive days.

SECONDARY OUTCOMES:
Change in workplace standing time at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  An activpal monitor will objectively assess habitual standing time for 24 hours over 7 consecutive days.
Change in workplace walking time at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  An activpal monitor will objectively assess habitual walking time for 24 hours over 7 consecutive days.
Change in whole day sitting time at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  An activpal monitor will objectively assess habitual sitting time for 24 hours over 7 consecutive days.
Change in whole day standing time at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  An activpal monitor will objectively assess habitual standing time for 24 hours over 7 consecutive days.
Change in whole day walking time at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  An activpal monitor will objectively assess habitual walking time for 24 hours over 7 consecutive days.
Change in body mass index at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from assessment of stature and body mass
Change in waist circumference at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from assessment of waist circumference
Change in hip circumference at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from assessment of hip circumference
Change in blood glucose at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from finger prick blood sampling
Change in blood cholesterol at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from finger prick blood sampling
Change in systolic blood pressure at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from automated blood pressure monitoring
Change in diastolic blood pressure at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from automated blood pressure monitoring
Change in endothelial function in the femoral artery at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from flow mediated dilation assessment
Change in musculoskeletal discomfort or pain: Self-reported using the Nordic Musculoskeletal Questionnaire | Baseline (week 0), 12 weeks, 9 months
  Discomfort or pain (neck, shoulders, elbows, wrist/hands, upper back, lower back, hips/thighs/buttocks, knees and ankles/feet) at 12 weeks and 9 months from baseline. The answer options are 'Yes' (discomfort or pain) or 'No' (no discomfort or pain - better outcome).
Change in wellbeing at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using the Short Form Health Survey v2 questionnaire. The answer options include scales from 'Excellent' (better outcome) to 'Poor', 'Yes limited a lot' to 'No not limited at all' (better outcome), and, 'All of the time' to 'None of the time' (better outcome).
Change in quality of life at 12 weeks and 9 months from baseline: EuroQol-5D | Baseline (week 0), 12 weeks, 9 months
  Self-reported using the EuroQol-5D questionnaire. The answer options include scales from 'I have no problems...' (better outcome) to 'I am unable to...', and, 'The worst health you can imagine' to 'The best health you can imagine' (better outcome).
Change in sleep at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using the Pittsburgh sleep quality index questionnaire. The answer options include scales from 'Not during the past month' (better outcome) to 'Three or more times a week', 'Very good' (better outcome) to 'Very bad', and, 'No problem at all' (better outcome) to 'A very big problem'.
Change in work engagement at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using the Utrecht Work Engagement scale. The answer options are scales from 'Never' to 'Always - everyday' (better outcome).
Change in occupational fatigue at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using the The Need for Recovery Scale. The answer options are 'Yes' or 'No'. The better outcome is question dependent.
Change in presenteeism at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using the Work Limitations Questionnaire. The answer options are scales from 'All of the time' to 'None of the time'. The better outcome is question dependent.
Change in subjective absenteeism at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using the Work Limitations Questionnaire. The answer options are scales from 'None' (better outcome) to '11 or more'.
Change in objective absenteeism at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from objectively assessed data to be provided from the participating organisation
Change in job satisfaction at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using a general job satisfaction questionnaire. The answer options are scales from 'Disagree strongly' to 'Agree strongly'. The better outcome is question dependent.
Change in work productivity at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Calculated from objectively assessed data to be provided from the participating organisation
Change in primary and secondary healthcare resource use at 12 weeks and 9 months from baseline | Baseline (week 0), 12 weeks, 9 months
  Self-reported using an adapted version of The Client Service Receipt Inventory questionnaire. The unit of measurement various across the questions with no scales.
Acceptability and feasibility of intervention components: Likert scale | 12 weeks and 9 months
  Self-reported by call agents using a Likert scale adapted from a previous trial. The answer options are scales from 'Very effective' (better outcome) to 'Very ineffective', and 'Strongly agree' (better outcome) to 'Strongly disagree'.
Acceptability and feasibility of the assessment protocol: Likert scale | 12 weeks and 9 months
  Self-reported by call agents using a Likert scale adapted from a previous trial. The answer options are scales from 'Strongly agree' (better outcome) to 'Strongly disagree'.
Acceptability and feasibility of the intervention components: Focus groups with call agents | 12 weeks and 9 months
  Call agents will take part in one focus group in which they will be asked to share their experiences and perceptions of the intervention components.
Acceptability and feasibility of the intervention components: Focus groups with team leaders | 12 weeks and 9 months
  Team leaders will take part in one focus group in which they will be asked to share their experiences and perceptions of the intervention components.
Acceptability and feasibility of the intervention components: Focus groups with middle managers | 12 weeks and 9 months
  Middle managers will take part in one focus group in which they will be asked to share their experiences and perceptions of the intervention components.
Acceptability and feasibility of the intervention components: Interview with senior managers | 12 weeks and 9 months
  Senior managers will take part in one interview in which they will be asked to share their experiences and perceptions of the intervention components.

CONTACTS AND LOCATIONS:
Overall Officials: Lee EF Graves, PhD, Principal Investigator — Liverpool John Moores University, Liverpool, Merseyside, United Kingdom, L3 2AT
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morris AS, Murphy RC, Hopkins ND, Low DA, Healy GN, Edwardson CL, Collins B, Timpson H, Shepherd SO, Cochrane M, Gavin D, Graves LEF. Sit Less and Move More-A Multicomponent Intervention With and Without Height-Adjustable Workstations in Contact Center Call Agents: A Pilot Randomized Controlled Trial. J Occup Environ Med. 2021 Jan 1;63(1):44-56. doi: 10.1097/JOM.0000000000002066. PMID 33122540